CLINICAL TRIAL: NCT04152720
Title: A Randomized, Multi-center, Open, Active-controlled Prospective Design Pilot Clinical Study to Evaluate the Efficacy and Safety of Prevention of Infection Foley Catheter as Compared to Conventional Foley Catheter in Patient Who Underwent Radical Cystectomy for Urological Disease
Brief Title: Evaluate the Efficacy and Safety of Prevention of Infection Foley Catheter as Compared to Conventional Foley Catheter
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Seoul National University Hospital (Other)
Collaborators: Seoul National University Bundang Hospital (Other); Samsung Medical Center (Other)
Responsible Party: Principal Investigator, Ja Hyeon Ku, Professor, Seoul National University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: APL_P_01
Record Dates: First submitted 2019-11-03; First posted 2019-11-05 (Actual); Last update posted 2019-11-05 (Actual); Status verified 2019-11

CONDITIONS: Urological Disease; Radical Cystectomy
Keywords: CAUTI; Catheter-associated urinary tract infection; Prevention of infection Foley Catheter
MeSH Terms: conditions — Urologic Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Prevention of infection Foley catheter (Active Comparator)
  Interventions: Device: Foley catheter
- Conventional Foley catheter (Active Comparator)
  Interventions: Device: Foley catheter

INTERVENTIONS:
Device: Foley catheter — If the subject is enrolled in this clinical trial, the test and control devices will be applied at baseline. All subjects will receive a urinary catheter at the site of the artificial bladder and the urethra after surgery, and temporary urinary replacement should be selected by the investigator at each institution in preparation for the possibility of postoperative blockage of the urinary catheter.
  After surgery, urine analysis and culture are performed on the 4th and 7th day, and urine analysis and culture are performed before the urethral catheter removal on the 14th (2 weeks) and the urethral catheter is removed. At this time, the urethral catheter tip is cut about 5-8 cm and cultured.

SUMMARY:
Comparison of effectiveness and safety of infection prevention silicone urinary catheters and conventional catheters for patients scheduled to perform urinary catheterization after radical cystectomy for urological diseases for more than 2 weeks Want to prove the clinical efficacy and safety.

ELIGIBILITY:
Inclusion Criteria:

1. Between 19 and 80 years old
2. Persons requiring urethral catheterization for more than 2 weeks after surgery * due to urological diseases

   * Radical cystectomy
3. Subjects who voluntarily decided to participate and signed the written informed consent
4. A person who can understand and follow the instructions and participate in the pre-clinical period.

Exclusion Criteria:

1. A person with a congenital abnormality in the urinary or reproductive system
2. Immunodeficiency disease (eg HIV infected)
3. Urinary tract fistula
4. Allergic history of the material used in the catheter
5. Symptomatic UTI by baseline time point
6. Dermatitis at the catheter insertion site
7. Pregnant or lactating women
8. A person who does not agree to contraceptive * in a medically accepted manner until the end of the study and 4 weeks after the end of the study.

   Medically acceptable contraceptive methods: condoms, oral contraceptives lasting at least 12 weeks, injectable or injectable contraceptives, intrauterine contraceptives, etc.
9. Inappropriate participation in the study, as determined by the investigator or investigator, as it may affect ethical or clinical trial results.
10. Patients on anti-thrombotic medication (excluding low-dose aspirin (100 mg, up to 300 mg / day))

Ages: 19 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Estimated)
Dates: Start 2018-08-03 (Actual); Primary Completion 2019-11-13 (Estimated); Study Completion 2020-03-30 (Estimated)

PRIMARY OUTCOMES:
1) Incidence of catheter-associated urinary tract infection (CAUTI) * 2 weeks after urethral catheterization | 2 weeks

SECONDARY OUTCOMES:
1) Period until catheter-associated urinary tract infection (CAUTI) occurs | 2 weeks
2) Incidence of Significant Bacterial Cultures in Urethral Catheter Tip Culture | 2 weeks
3) Catheter related complication rate | 2 weeks
4) Catheter-associated urinary tract infection 2 weeks after urethral catheter insertion in test and control groups | 2 weeks
5) Antibiotic administration period due to catheter-related urinary tract infection | 2 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Seoul National University Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: Undecided